CLINICAL TRIAL: NCT01021670
Title: A Prospective, Observational Study of Men With Premature Ejaculation Who Are Treated With PRILIGY or Alternate Care
Brief Title: An Observational Study of Men With Premature Ejaculation Who Are Treated With Dapoxetine Hydrochloride or Alternate Care Defined as Any Treatment Other Than Dapoxetine Hydrochloride
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016477; The PAUSE Study (Other: Janssen Research & Development, LLC); R096769PRE4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Sexual Dysfunction, Physiological; Ejaculation
Keywords: Dapoxetine hydrochloride; Priligy; Premature ejaculation; Non-dapoxetine hydrochloride treatment(s)
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Premature Ejaculation | interventions — dapoxetine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 001: Dapoxetine hydrochloride One 30 mg tablet up to a maximum of one 60 mg tablet approximately 1 to 3 hours prior to prior to sexual activity once every 24 hours as needed for 12 weeks
  Interventions: Drug: Dapoxetine hydrochloride
- 002: Alternate care/non-dapoxetine hydrochloride treatment(s) As prescribed or directed
  Interventions: Other: Alternate care/non-dapoxetine hydrochloride treatment(s)

INTERVENTIONS:
Drug: Dapoxetine hydrochloride — One 30 mg tablet up to a maximum of one 60 mg tablet approximately 1 to 3 hours prior to prior to sexual activity once every 24 hours as needed for 12 weeks
  Groups: 001
Other: Alternate care/non-dapoxetine hydrochloride treatment(s) — As prescribed or directed
  Groups: 002

SUMMARY:
The purpose of the study is to collect information regarding the safety of dapoxetine hydrochloride when used in clinical practice to treat men with premature ejaculation. Dapoxetine hydrochloride is a selective inhibitor of serotonin reuptake that is indicated for the treatment of patients with premature ejaculation.

DETAILED DESCRIPTION:
This is a 12-week, observational study to collect and evaluate safety data for dapoxetine hydrochloride and alternate care/non-dapoxetine hydrochloride treatment(s) defined as any treatment (eg, oral, topical, or behavioral) other than dapoxetine hydrochloride, which have been recommended and prescribed for men who have a diagnosis of premature ejaculation. The primary objective of the study is to describe the safety profile of dapoxetine hydrochloride when used in clinical practice. The safety of dapoxetine hydrochloride will be assessed duing the study by monitoring the occurrence of all adverse events experienced by patients including adverse events of special interest (eg, syncope, characterized as loss of consciousness). Safety will also be assessed by monitoring patient use of all concomitant medications/treatments including prescription medications, over the counter medications, vitamins and herbal supplements, and other types of therapies such as electrical stimulation, acupuncture, special diets, and exercise regimens. Approximately 12,000 men with premature ejaculation will be enrolled in the study of which approximately 6,000 patients will be treated with dapoxetine hydrochloride. All patients who present to the practice for an evaluation of premature ejaculation, or who have a diagnosis of premature ejaculation and are currently being treated will be considered for enrollment in the study. All treatment decisions will be made at the discretion of the participating health care provider. The study will consist of 3 periods: a pre-observational (screening/baseline) period (Visit 1), an 12-week observational period (Visits 2, 3, and 4), and a 4-week post-observational period. At Visit 1, the health care provider will make or confirm the diagnosis of premature ejaculation and determine if treatment with dapoxetine hydrochloride or alternate care/non-dapoxetine hydrochloride is appropriate for the patient. There will be no study-specific selection criteria other than the guidance provided by the Summary of Product Characteristics for dapoxetine hydrochloride as it is intended that the participating health care provider will use the Summary of Product Characteristics for dapoxetine hydrochloride as a guide to identify appropriate patients for the study, and the types of patients who should use caution or avoid using dapoxetine hydrochloride. If the healthcare provider determines that the patient is a candidate for the study, he/she will explain the details of the study to the patient. Patients who are interested in participating in the study should be willing and able to be treated with dapoxetine hydrochloride and to continue to participate in the study as long as dapoxetine hydrochloride continues to be administered for the duration of the 12-week observational period, even in those situations where topical and/or behavioral alternate care treatments are added to the dapoxetine hydrochloride treatment regimen. Patients who wish to participate in the study will be asked to sign and date an informed consent to allow the health care provider to collect information required for the study. At Visit 1, a signed informed consent form will be obtained from the patient and information will be collected including demographics (for example, the patient's race and age), medical history including premature ejaculation history, physical examination findings, and orthostatic vital sign (blood pressure and heart rate/pulse) measurements. If the health care provider determines that the patient should be treated with dapoxetine hydrochloride, the health care provider will instruct the patient on the administration of dapoxetine hydrochloride according to the dosage and administration guidelines in the Summary of Product Characteristics for dapoxetine hydrochloride as follows: the recommended starting dose of dapoxetine hydrochloride is 30 mg, taken with or without food with at least one full glass of water approximately 1 to 3 hours prior to prior to sexual activity once every 24 hours as needed. If the effect of dapoxetin hydrochloride at a dose of 30 mg is insufficient and the side effects are acceptable, the dose may be increased to the maximum recommended dose of 60 mg. If the health care provider determines that the patient should be treated with alternate care/non-dapoxetine hydrochloride treatment(s), the health care provider will instruct the patient on the administration of those treatments as prescribed or directed. Following Visit 1, all patients will participate in a 12-week observational period where they will return for up to 3 study visits (Visits 2, 3, and 4) according to the health care provider's local practice. At each visit, the health care provider will evaluate if the dose of dapoxetine hydrochloride or alternate care/non-dapoxetine hydrochloride treatment(s) needs to be increased or decreased and information regarding the occurrence of adverse events and the use of concomitant medications/treatment will be collected. Approximately 4 weeks following the end of the 12-week observational period or the patient's last visit in the study, the health care provider will contact the patient by telephone to assess the occurrence of any adverse events experienced by the patient and the use of any concomitant medications or treatments taken since the last study visit. Additional telephone contact with the patient may be performed by the health care provider to obtain additional information to determine the patient's safety or survival status. Regardless of the patient's status at the end of the study (ie, completed, discontinued treatment, withdrew early), patients who receive dapoxetine hydrochloride will be asked to complete a survey to provide feedback to the healthcare provider on the whether or not the dapoxetine hydrochloride Patient Brochure and/or Patient Information Leaflet was useful and informative. Patients may only participate in the study one time. Patients who receive dapoxetine hydrochloride in the study should not be enrolled again to receive alternate care/non-dapoxetine hydrochloride treatment(s) upon study completion or discontinuation of dapoxetine hydrochloride). The recommended starting dose of dapoxetine hydrochloride is 30 mg, taken with or without food with at least 1 full glass of water approximately 1 to 3 hours prior to prior to sexual activity once every 24 hours as needed. Patients will take dapoxetine hydrochloride for 12 weeks during the observational period of the study. Alternate care/non dapoxetine hydrochloride treatment(s) will be administered to patients in accordance with the prescribing information and/or directions for use.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the therapeutic indication stated in the Summary of Product Characteristics for dapoxetine hydrochloride, patients will be candidates for enrollment if they have an intravaginal ejaculatory latency time of less than two minutes
* Persistent or recurrent ejaculation with minimal sexual stimulation before, on, or shortly after penetration and before the patient wishes
* Marked personal distress or interpersonal difficulty as a consequence of premature ejaculation
* Poor control over ejaculation

Exclusion Criteria:

* In accordance with the contraindications, special warnings and precautions for use as stated in the Summary of Product Characteristics for dapoxetine hydrochloride, patients will be excluded from treatment if they have hypersensitivity to dapoxetine hydrochloride or to any of the excipients
* Significant pathological cardiac conditions such as: heart failure (New York Heart Association [NYHA] class II-IV), conduction abnormalities (second or third degree atrioventicular (AV) block or sick sinus syndrome) not treated with a permanent pacemaker, significant ischemic heart disease, or significant valvular disease
* Concomitant treatment with monoamine oxidase inhibitors (MAOIs), or within 14 days of discontinuing treatment with an MAOI
* Concomitant treatment with thioridazine, concomitant treatment with serotonin reuptake inhibitors (selective serotonin reuptake inhibitors [SSRIs], serotonin-norepinephrine reuptake inhibitors [SNRIs], tricyclic antidepressants [TCAs)] or other medicinal/herbal products with serotonergic effects (for example, L-tryptophan, triptans, tramadol, linezolid, lithium, St. John's Wort (Hypericum perforatum)
* Concomitant treatment of potent CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, saquinavir, telithromycin, nefazadone, nelfinavir, atazanavir, etc.
* Moderate and severe hepatic impairment

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men diagnosed with premature ejaculation will be enrolled in the study by participating health care providers in clinical practice settings.
Sampling Method: Non-Probability Sample
Enrollment: 10027 (Actual)
Dates: Start 2009-09; Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is safety. Safety will be assessed by monitoring the occurrence of adverse events and the use of concomitant medications or therapies during the study. | Safety will be assessed at Visit 1 through 4 during the 12 week observation period and up to approximately 4 weeks after the End-of-Observation/Early Withdrawal Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (212):
- Austria (3):
  - Karpfenberg
  - Reutte
  - Vienna
- Finland (5):
  - Helsinki
  - Kouvola
  - Mikkeli
  - Oulu
  - Turku
- Germany (113):
  - Ahlen
  - Ahrensburg
  - Apolda
  - Bad Doberan
  - Bad Schönborn
  - Bamberg
  - Bautzen
  - Berlin
  - Bonn
  - Böblingen
  - Braunschweig
  - Bremen
  - Bruchsal
  - Castrop-Rauxel
  - Celle
  - Chemnitz
  - Cologne
  - Dachau
  - Dessau
  - Dorsten
  - Dortmund
  - Dossenheim
  - Dresden
  - Duisburg
  - Düren
  - Düsseldorf
  - Eisenberg
  - Eisleben Lutherstadt
  - Erfurt
  - Erlangen
  - Essen
  - Frankfurt
  - Garmisch-Partenkirchen
  - Gotha
  - Göppingen
  - Grimma
  - Grünstadt
  - Hagenow
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Heilbronn
  - Hemmoor
  - Herford
  - Herten
  - Herzogenaurach
  - Höchberg
  - Höchheim
  - Jena
  - Kaiserslautern
  - Karlsruhe
  - Kempten
  - Kiel
  - Kirchheim
  - Kleinmachnow
  - Krefeld
  - Kronach
  - Lampertheim
  - Landsberg
  - Leipzig
  - Leverkusen
  - Lichtenfels
  - Lüdinghausen
  - Magdeburg
  - Markkleeberg
  - Mülheim
  - München
  - Münster
  - Neckargemünd
  - Neu-Ulm
  - Neumünster
  - Neuss
  - Nordhausen
  - Nuremberg
  - Oberursel
  - Oranienburg
  - Osnabrück
  - Ostfildern
  - Peine
  - Planegg
  - Plauen
  - Radebeul
  - Rastatt
  - Remscheid
  - Reutlingen
  - Rinteln
  - Rostock
  - Rottenberg
  - Rottweil
  - Sangerhausen
  - Schleswig
  - Schriesheim
  - Schwerin
  - Senftenberg
  - Sindelfingen
  - Sömmerda
  - Speyer
  - Stadthagen
  - Starnberg
  - Strausberg
  - Stuttgart
  - Taucha
  - Ulm
  - Unterschleissheim
  - Velbert
  - Villingen-Schwenningen
  - Wiesbaden
  - Wiesloch
  - Wolfenbüttel
  - Wolfsburg
  - Wuppertal
  - Zwickau
- Portugal (10):
  - Aveiro
  - Braga
  - Castelo Viegas
  - Estoril
  - Lisbon
  - Matosinhos Municipality
  - P-1100 Lisboa N/A
  - Portimão
  - Póvoa Do Varzim
  - Santo Tirso
- Spain (73):
  - A Coruña
  - Alcorcón
  - Alginet
  - Alicante
  - Almería
  - Aravaca
  - Avilés
  - Badalona
  - Barakaldo
  - Barcelona
  - Burgos
  - Cadiz
  - Calatayud
  - Calella
  - Castellon
  - Ciudad Real
  - Córdoba
  - Cullera
  - Donostia / San Sebastian
  - el Prat de Llobregat
  - Gandia
  - Girona
  - Granada
  - Ibiza Town
  - Jaén
  - L'Hospitalet de Llobregat
  - Las Palmas de Gran Canaria
  - León
  - Llanera
  - Lleida
  - Logroño
  - Los Boliches
  - Lugo
  - Madrid
  - Manacor
  - Marbella
  - Mataró
  - Málaga
  - Murcia
  - Ontiyent
  - Ourense
  - Oviedo
  - Palamós
  - Palma de Mallorca
  - Pamplona
  - Parla
  - Pontevedra
  - Port de Bollenca
  - Requena
  - Ribeira
  - Rota
  - Sabadell
  - Salamanca
  - San Cristóbal de La Laguna
  - San Sebastián de los Reyes
  - Sanlúcar de Barrameda
  - Sant Joan d'Alacant
  - Santa Cruz de Tenerife
  - Santander
  - Santiago de Compostela
  - Seville
  - Silla
  - Tarragona
  - Terrassa
  - Toledo
  - Utrera
  - Valencia
  - Valladolid
  - Vigo
  - Vilanova i la Geltrú
  - Villamayor
  - Xátiva
  - Zaragoza
- Sweden (8):
  - Billdal
  - Eskilstuna
  - Gothenburg
  - Karlshamn
  - Luleå
  - Lund
  - Motala
  - Stockholm

REFERENCES:
- See also: A Prospective, Observational Study of Men With Premature Ejaculation Who Are Treated With PRILIGY™ or Alternate Care — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=820&filename=CR016477_CSR.pdf